CLINICAL TRIAL: NCT01526447
Title: Effects of Craniosacral Therapy on Chronic Neck Pain: A Randomized Controlled Trial
Brief Title: Effects of Craniosacral Therapy on Chronic Neck Pain
Acronym: CranioS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, Postdoctoral Research Fellow, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-4850
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Neck Pain
Keywords: Neck Pain; Craniosacral Manipulation; Complementary Therapies; Randomized Controlled Trial; Sensory Thresholds; Quality of Life
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Craniosacral Therapy (CST) (Experimental): Each participant of the experimental group receives 8 Craniosacral Therapy units once a week of 45 minutes.
  Interventions: Procedure: Craniosacral Therapy
- Sham Craniosacral Therapy (SHAM) (Sham Comparator): Each participant of the sham group receives 8 sham therapy units once a week of 45 minutes.
  Interventions: Procedure: Sham Craniosacral Therapy

INTERVENTIONS:
Procedure: Craniosacral Therapy — Standardized therapy protocol (according to Upledger): Still point technique, diaphragm release, compression-decompression and lift techniques of the cranial bones, facial balancing in the region of shoulder and pelvis and somato-emotional unwinding
  Arms: Craniosacral Therapy (CST)
Procedure: Sham Craniosacral Therapy — Standardized sham protocol: Placing hands on various parts of the clothed body for two minutes each time without therapeutic intention
  Arms: Sham Craniosacral Therapy (SHAM)

SUMMARY:
The purpose of this randomized controlled trial is to determinate the efficacy and safety of Craniosacral Therapy in the treatment of chronic unspecific neck pain.

DETAILED DESCRIPTION:
Craniosacral Therapy (CST) is a variation of osteopathic manipulation with an integrative approach. By soft manual palpation of the craniosacral and fascia system sensory, motor, cognitive, and emotional processes can be influenced. In the prevention and treatment of chronic pain syndromes Craniosacral Therapy is demonstrated to be effective in clinical practice and quite a few scientific trials. But yet there are no randomized controlled studies concerning to chronic neck pain. So the aim of this study is to investigate whether a total of 8 CST units of 45 minutes will be effective in patients suffering from chronic nonspecific neck pain in contrast to sham therapy of the same extent. The prospective study design includes measurement points at baseline, post treatment, and 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Chronic unspecific neck pain for at least 3 months
* Mean neck pain of moderate intensity (>/=45mm on VAS)
* Therapy-naive subjects

Exclusion Criteria:

* Specific neck pain due to severe deformity of the spine, prolapse, rheumatic or neurological disorder, trauma, operation or cancer
* other severe somatic or psychiatric comorbidity
* pregnancy
* regular intake of opiates, corticosteroids (>10mg prednisolon), muscle relaxants or antidepressants
* recent invasive or manipulative treatment of the spine
* participation in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain intensity | week 8
  Pain intensity on a 100mm visual analogue scale (VAS)

SECONDARY OUTCOMES:
Pain intensity in motion | week 8
  Pain intensity induced by flexion, extension, lateral flexion and rotation of the head on a 100mm visual analogue scale (VAS)
Pressure pain threshold | week 8
  Pressure pain threshold (PPT) measured with an algometer on predefined muscles and the pain maximum
Disability | week 8
  Measured by the Neck Disability Indx (NDI)
Quality of life | week 8
  Measured by the Short-Form Health Survey (SF-12)
Well being | week 8
  Measured by the Questionnaire for Assessing Subjective Physical Well-Being (FEW-16)
Anxiety and depression | week 8
  Measured by the Hospital Anxiety and Depression Scale (HADS)
Stress perception | week 8
  Measured by the Perceived Stress Questionnaire (PSQ-20)
Pain acceptance | week 8
  Measured by the Emotional and Rational Disease Acceptance Questionnaire (ERDA)
Body awareness | week 8
  Measured by the Scale of Body Connection (SBC)
Global Impression | week 8
  Measured by the Patient Global Impression of Improvement Questionnaire (PGI-I)
Safety | week 8
  All adverse events are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Director — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University Duisburg-Essen, Germany
Locations (1):
- Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Haller H, Ostermann T, Lauche R, Cramer H, Dobos G. Credibility of a comparative sham control intervention for Craniosacral Therapy in patients with chronic neck pain. Complement Ther Med. 2014 Dec;22(6):1053-9. doi: 10.1016/j.ctim.2014.09.007. Epub 2014 Oct 6. PMID 25453528
- [Result] Haller H, Lauche R, Cramer H, Rampp T, Saha FJ, Ostermann T, Dobos G. Craniosacral Therapy for the Treatment of Chronic Neck Pain: A Randomized Sham-controlled Trial. Clin J Pain. 2016 May;32(5):441-9. doi: 10.1097/AJP.0000000000000290. PMID 26340656